CLINICAL TRIAL: NCT05178134
Title: A Phase 2 Immunological Bridging Study Assessing the Non-inferiority of a New Formulation of ETVAX®. A Prospective Double-blind, Randomized Study in Healthy Volunteers.
Brief Title: A Phase 2 Bridging Study to Assess the New Formulation of ETVAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scandinavian Biopharma AB (Industry)
Collaborators: Göteborg University (Other); Aurevia (Industry); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OEV-125; 2021-001541-13 (EudraCT Number)
Record Dates: First submitted 2021-12-03; First posted 2022-01-05 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healty Volunteers; Preventable Disease, Vaccine
Keywords: Prophylaxis against diarrhea due to enterotoxigenic E. coli
MeSH Terms: conditions — Vaccine-Preventable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Other parts will be blinded except unblinded person who prepares the doses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The wet formulation of ETVAX. (Active Comparator): The wet formulation consists of a liquid suspension of inactivated bacteria (ETEX 21-24) and LCTBA in one vial, freeze-dried dmLT adjuvant in a second vial, and effervescent buffer granules in a separate sachet. Prior to administration, the buffer is dissolved in 150 ml tap water, followed by the addition of the content of the vaccine vial (inactivated bacteria mixed with LCTBA) and reconstituted and diluted adjuvant dmLT from the second vial.
  Interventions: Biological: Etvax
- The partially dried formulation of selected components of ETVAX. (Active Comparator): The partially dried formulation, dmLT and LCTBA are spray-dried and mixed with the buffer granules and stabilizing excipients in a sachet. Prior to administration, the content of the buffer sachet (buffer, dmLT, and LCTBA) is dissolved in 150 ml tap water, followed by the addition of a liquid suspension of inactivated bacteria (ETEX 21-24).
  Interventions: Biological: Etvax

INTERVENTIONS:
Biological: Etvax — Preparation of complete Wet formulation. The vaccine supplied as a liquid, is mixed with the 150 ml of sodium bicarbonate buffer solution on the day of preparation for use on dosing day.
  Just prior to administration 10 µg of dmLT is added by pipette (50 µl).
  Arms: The wet formulation of ETVAX.
Biological: Etvax — Preparation of partially dry formulation. The partially dry formulation of vaccine is prepared by adding the effervescent powder containing the dmLT and LCTBA to 150 ml of water. After mixing, the content of the vaccine vial is added to the mixture and the vaccine is administered to the volunteer within 30 minutes after adding the buffer powder to the water.
  Arms: The partially dried formulation of selected components of ETVAX.

SUMMARY:
This is a phase 2,prospective double-blind, randomized, parallel-group study with the aim to demonstrate non-inferiority, in terms of immunogenicity, between the wet formulation and a newly developed partially dried formulation of selected components of ETVAX.

DETAILED DESCRIPTION:
This is a phase 2, prospective double-blind, randomized, parallel-group study with the aim to demonstrate non-inferiority, in terms of immunogenicity, between the wet formulation and a newly developed partially dried formulation of selected components of ETVAX. A total number of 126 subjects is planned to be included in each arm of the study, i.e. 252 subjects in total. Assuming a 10% dropout rate the target number of subjects to be recruited per study arm is therefore 140, i.e. 280 subjects in total. Healthy volunteers between 18-50 years will be eligible for enrolment into the study.

Eligible subjects will be randomized on Day 1 (Visit 2) to receive either of the two oral formulations of ETVAX (1:1) and consecutively included the study. The treatment allocation (Wet formulation/Partially dried formulation) will be double-blind. The study subjects will receive two oral doses, two weeks apart (Day 1/Visit 2 and Day 15 /Visit 3).The dosing will occur at the clinic (CTC in Gothenburg, Sweden). A follow-up visit will be performed 7 days after the last (second) dose in all study subjects

The primary endpoint to be measured for each patient in the study is response (yes/no) to a vaccine. A vaccine responder will be defined by a ≥2-fold increase in IgA and/or IgG antibody levels against LTB in serum between post- compared to pre-immunization samples. The response rates (seroconversion rates) of IgA and/or IgG anti-LTB antibodies in serum will be derived and compared between the two treatment groups.

The secondary endpoint to be measured for each patient in the study is the occurrence of solicited symptoms for six days after each vaccination (day of vaccination and five subsequent days).

Exploratory analyses will be done to evaluate if ETVAX vaccination induces circulating antigen specific memory B- and/or T cells that can be assessed using recently established laboratory assays.

For the exploratory analyses, subgroups of subjects (n=20-40, evenly distributed between the two treatment arms) will participate in additional follow-up visits 5± 1, 30± 7 and 90± 14 days after the second dose. Blood samples will be collected on all exploratory visits. The extra visits and analyses for exploratory analyses may continue after the main part of the study has been completed and the database locked.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-50 years, inclusive at the time of signing the informed consent.
* Healthy constitution as established by medical history and physical examination.
* Willing and able to give written informed consent for participation in the study.
* Able to comply with study activities, as judged by the Investigator.
* Female Participants:
* Women of child-bearing potential (for definition see Section 9.3.6 in the protocol):
* Have to agree to use an acceptable birth control method during participation in the investigation (see Section 9.3.6).
* A negative pregnancy test (beta human chorionic gonadotropin dipstick test in urine) at Visit 2/Day 1 will be required.
* Male Participants:
* Have to agree to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined in Section 9.3.6

Exclusion criteria

* An acute or chronic medical condition that, in the opinion of the investigator/physician, would render ingestion of the investigational products unsafe or would interfere with the evaluation of responses. This includes, but is not limited to gastrointestinal diseases, and autoimmune diseases.
* Current malignancy or history of malignancy during the last five years, based on anamnesis.
* Gastroenteritis within two weeks prior to vaccination.
* Regular use of laxatives, antacids or other agents that lower stomach acidity.
* Any planned major surgery during the duration of the study.
* After 10 minutes supine rest, any vital signs outside the following ranges:
* Systolic BP > 160 mm Hg
* Diastolic BP > 100 mm Hg
* Heart rate < 40 or >85 beats per minute
* Antibiotic therapy within two weeks prior to the vaccination.
* Known Hepatitis A, B, C, and/or HIV infection.
* Concomitant intake of immunomodulating drugs during the study period or less than 3 months prior to the first immunization, with the following exceptions: oral anti-histamines are not allowed during the study period or less than 3 weeks prior to the first immunization. Local anti-histamine treatment is allowed during the study period.
* Any other significant medical conditions (e.g. poorly controlled psychiatric condition) judged by the Investigator to preclude entry.
* Intends to receive any other vaccine during the study period, or within two weeks prior to trial vaccination.
* Has previously received Dukoral or any type of ETEC or cholera vaccines.
* Brought up in ETEC-endemic areas (e.g., urban and rural areas of Central and South America, Caribbean, most countries in Asia, Africa, etc.).
* Has travelled to ETEC-endemic areas within the last 3 years OR spent > two months in ETEC endemic areas during the last 10 years.
* Intends to travel to ETEC endemic countries during the study period.
* Known or suspected history of drug, chemical or alcohol abuse, as deemed by the investigator/physician.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to ETVAX®.
* Participation in any other clinical study that included drug treatment with the last administration within the past 3 months prior to administration of study treatment in this study. Patients consented and screened but not dosed in previous clinical studies are not excluded.
* Concomitant participation in any other clinical study.
* Females who are pregnant as determined by urine test at inclusion and prior to each vaccination.
* Females who are nursing.
* Unable to participate in all study visits.
* Any condition or circumstance which would make the subject unsuitable for participation in the study in the opinion of the investigator/physician.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Curiac, MD, Principal Investigator — Clinical Trial Center, CTC, Gothia Forum
Locations (1):
- Clinical Trial Center, CTC, Gothenburg, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- The Wet Formulation of ETVAX.: The wet formulation consists of a liquid suspension of inactivated bacteria (ETEX 21-24) and LCTBA in one vial, freeze-dried dmLT adjuvant in a second vial, and effervescent buffer granules in a separate sachet. Prior to administration, the buffer is dissolved in 150 ml tap water, followed by the addition of the content of the vaccine vial (inactivated bacteria mixed with LCTBA) and reconstituted and diluted adjuvant dmLT from the second vial.
  Etvax: Preparation of complete Wet formulation. The vaccine supplied as a liquid, is mixed with the 150 ml of sodium bicarbonate buffer solution on the day of preparation for use on dosing day.
  Just prior to administration 10 µg of dmLT is added by pipette (50 µl).
Period: Overall Study
Arm/Group | The Wet Formulation of ETVAX. | The Partially Dried Formulation of Selected Components of ETVAX.
Started | 140 | 140
Completed | 139 | 139
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Wet Formulation of ETVAX. | The Partially Dried Formulation of Selected Components of ETVAX. | Total
Number analyzed (Participants) | 140 | 140 | 280
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.0 (9.70) | 32.2 (9.54) | 31.6 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 87 | 173
  Male | 54 | 53 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 139 | 139 | 278
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 140 | 140 | 280

OUTCOME MEASURES:

1. Primary Outcome: Vaccine Response
Description: The primary endpoint to be measured for each patient in the study is response (yes/no) to a vaccine. A vaccine responder will be defined by a ≥2-fold increase in IgA and/or IgG antibody levels against LTB in serum between post- compared to pre-immunization samples. The response rates (seroconversion rates) of IgA and/or IgG anti-LTB antibodies in serum will be derived and compared between the two treatment groups.
Time Frame: 3 weeks
Population: Per Protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | The Wet Formulation of ETVAX. | The Partially Dried Formulation of Selected Components of ETVAX.
Number analyzed (Participants) | 137 | 133
Participants | 116 | 110
Statistical Analysis 1: Comparison: The Wet Formulation of ETVAX. vs The Partially Dried Formulation of Selected Components of ETVAX; Test type: Non-Inferiority — Non-inferiority margin was set to -15% (on an absolute scale); Difference in response rates = -0.020, 95% CI 2-sided [-0.108 to 0.069]

2. Secondary Outcome: Solicited Symptoms After Vaccination
Description: Occurrence of solicited symptoms for six days after each vaccination (day of vaccination and five subsequent days).
Time Frame: 3 weeks
Population: 140 subjects in each group received one vaccine dose and 139 subjects in each group received two vaccine doses.
Measure: Count of Participants; unit: Participants
Arm/Group | The Wet Formulation of ETVAX. | The Partially Dried Formulation of Selected Components of ETVAX.
Number analyzed (Participants) | 140 | 140
Participants
  Subjects who experienced solicited AEs within 6 days after first dose: Abdominal pain | 23 | 22
  Subjects who experienced solicited AEs within 6 days after first dose: Nausea | 17 | 20
  Subjects who experienced solicited AEs within 6 days after first dose: Vomiting | 3 | 3
  Subjects who experienced solicited AEs within 6 days after first dose: Loose stools/Diarrhea | 24 | 33
  Subjects who experienced solicited AEs within 6 days after first dose: Fever | 3 | 0
  Subjects who experienced solicited AEs within 6 days after first dose: No solicited symptom | 70 | 62
  Subjects who experienced solicited AEs within 6 days after second dose: number analyzed (Participants) | 139 | 139
  Subjects who experienced solicited AEs within 6 days after second dose: Abdominal pain | 24 | 12
  Subjects who experienced solicited AEs within 6 days after second dose: Nausea | 22 | 20
  Subjects who experienced solicited AEs within 6 days after second dose: Vomiting | 4 | 5
  Subjects who experienced solicited AEs within 6 days after second dose: Loose stools/Diarrhea | 27 | 24
  Subjects who experienced solicited AEs within 6 days after second dose: Fever | 3 | 0
  Subjects who experienced solicited AEs within 6 days after second dose: No solicited symptom | 59 | 78

3. Other Pre Specified Outcome: Levels of IgA and IgG Antibodies Mononuclear Cells (PBMCs)
Description: Evaluation if ETVAX® vaccination induces circulating antigen specific memory B- and/or T cells.
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Collection of unsolicited AEs started with the first intervention with the study vaccine and continued until the last follow-up assessment 7 days (6-10 days) after study vaccine dose 2.
Description: Collection of Adverse Events:
  * Diary solicited: Registration of solicited symptoms for 6 days after each vaccination through a diary where questions about solicited symptoms were included. The occurrence of solicited symptoms for 6 days after each vaccination was defined as secondary outcome measure in this study.
  * Other: Unsolicited adverse events where the collection was not primarily through diaries. The collection period for unsolicited adverse events was the entire study period.
Arm/Group | The Wet Formulation of ETVAX. | The Partially Dried Formulation of Selected Components of ETVAX.
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/140
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/140
Other Adverse Events (participants affected / at risk) | 107/140 | 102/140
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Wet Formulation of ETVAX. (N=140) | The Partially Dried Formulation of Selected Components of ETVAX. (N=140)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Inner ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 19 (21) | 14 (18)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 7 (8) | 5 (5)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Hunger (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes Simplex (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 12 (12) | 11 (13)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Otosalpingitis (Infections and infestations) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Papilloma conjunctival (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4)
Exertional headache (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 43 (59) | 40 (55)
Migraine (Nervous system disorders) | 1 (2) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 13 (14) | 5 (5)
Premenstrual dysphoric disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 36 (62) | 30 (38)
Diarrhoea (Gastrointestinal disorders) | 41 (67) | 42 (71)
Nausea (Gastrointestinal disorders) | 32 (47) | 33 (46)
Pyrexia (General disorders) | 7 (7) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (8) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT05178134/Prot_SAP_000.pdf